CLINICAL TRIAL: NCT03653715
Title: Clinical Performance Study of Clerio Single Vision and Bifocal Contact Lens Designs Immediately Following Insertion
Brief Title: Bifocal Contact Lens Study for Adults With Age-Related Near Vision Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clerio Vision, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CVR-18-001
Record Dates: First submitted 2018-08-27; First posted 2018-08-31 (Actual); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Presbyopia
Keywords: Refractive Errors; Myopia; Hyperopia; Astigmatism
MeSH Terms: conditions — Presbyopia; Refractive Errors; Myopia; Hyperopia; Astigmatism

STUDY DESIGN:
Intervention Model Description: This single center study is a device feasibility, two-arm, double-masked (participants and outcomes assessor), repeated measures, cross-sectional design. Each participant is tested with the four (4) study devices (i.e., contact lenses), one (1) test lens and three (3) control lenses, in randomized order. Participants are masked to each lens they wear.
Who Masked: Participant, Outcomes Assessor
Masking Description: The Principal Investigator and Clinical Research Technicians, because they handle the contact lenses both in and out of their packaging, are not masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Test Device (Experimental): Within this arm the Clerio Vision LIRIC-modified Bifocal Contact Lens is administered.
  Interventions: Device: Clerio Vision LIRIC-modified Bifocal Contact Lens
- Control Devices (Active Comparator): Within this arm the Johnson & Johnson 1-Day Acuvue Moist Multifocal Contact Lens, Johnson & Johnson 1-Day Acuvue Moist Contact Lens, and Clerio Vision Single Vision Contact Lens are administered.
  Interventions: Device: Johnson & Johnson 1-Day Acuvue Moist Multifocal Contact Lens; Device: Johnson & Johnson 1-Day Acuvue Moist Contact Lens; Device: Clerio Vision Single Vision Contact Lens

INTERVENTIONS:
Device: Clerio Vision LIRIC-modified Bifocal Contact Lens — Within this arm the investigational acofilcon B material bifocal contact lens, which has been modified with the laser and is the focus of the study, is tested. This lens is one of four (4) administered to each participant, tested on either visit 2 or 3 according to the randomization schedule, for a period of approximately 20 minutes.
  Other Names: Clerio Vision Bifocal Contact Lens; Clerio Vision Multifocal Contact Lens; Laser-Induced Refractive Index Change (LIRIC) Bifocal Contact Lens
  Arms: Test Device
Device: Johnson & Johnson 1-Day Acuvue Moist Multifocal Contact Lens — Within this arm the control etafilcon A material bifocal contact lens, which is commercially available, is tested. This lens is one of four (4) administered to each participant, tested on either visit 2 or 3 according to the randomization schedule, for a period of approximately 20 minutes.
  Other Names: Commercially Available Multifocal Contact Lens; Control Multifocal Contact Lens; Etafilcon A
  Arms: Control Devices
Device: Johnson & Johnson 1-Day Acuvue Moist Contact Lens — Within this arm the control etafilcon A material single vision contact lens, which is commercially available, is tested. This lens is one of four (4) administered to each participant, tested on either visit 2 or 3 according to the randomization schedule, for a period of approximately 20 minutes.
  Other Names: Commercially Available Single Vision Contact Lens; Control Single Vision Contact Lens; Etafilcon A
  Arms: Control Devices
Device: Clerio Vision Single Vision Contact Lens — Within this arm the control acofilcon B material single vision contact lens, the material of which is commercially available from Contamac Ltd, is tested. This lens is one of four (4) administered to each participant, tested on either visit 2 or 3 according to the randomization schedule, for a period of approximately 20 minutes.
  Other Names: Contamac 49 Single Vision Contact Lens; Control Single Vision Contact Lens; Acofilcon B
  Arms: Control Devices

SUMMARY:
The primary objective of this study is to evaluate the distance, intermediate and near visual performance of Clerio designed single vision and Clerio designed LIRIC modified bifocal lenses (+2.00D add) compared to commercially available single vision and multifocal lenses.

DETAILED DESCRIPTION:
Clerio Vision Inc. has licensed a new femtosecond based laser procedure discovered by researchers at the University of Rochester known as Laser Induced Refractive Index Customization (LIRIC), which allows the alteration of the optical design of a finished soft hydrogel contact lens. Clerio Vision Inc. scientists have developed a diffractive multifocal optical design using the LIRIC procedure which shows an increase of the depth of focus of the contact lens when measured on an optical bench. It is hypothesized that a presbyopic patient wearing a soft contact lens of this design will experience an improvement in intermediate and near vision over that provided by their distance corrected single vision contact lenses, without significantly impacting their distance vision. The purpose of this feasibility study is the on-eye evaluation of the performance of the Clerio Vision designed and LIRIC modified soft contact lenses. Results from this study will guide future development of these potential products.

ELIGIBILITY:
Inclusion Criteria:

* Legal age (at least 21) on the date the Informed Consent Form (ICF) is signed and have the capacity to provide voluntary informed consent
* Able to read, understand and provide written informed consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved ICF and provide authorization as appropriate for local privacy regulations.
* Willing and able to comply with all study instructions/procedures.
* Best Distance Spherical Corrected Visual Acuity (BDSCVA) in at least one eye of 20/25 (0.10 logMAR).
* Physiologically normal anterior segments not exhibiting clinically significant biomicroscopy findings.
* Previous experience with contact lenses.
* Distance spectacle spherical correction in at least one eye within +/- 5D of the study lens power (-3.00D).
* Habitual spectacle addition (at 40cm) of at least +1.00D.
* Refractive astigmatism less than -2.75D.
* Most recent complete eye examination was within the last 24 months of the date of study completion.

Exclusion Criteria:

* Currently participating in any drug or device clinical investigation during the period of study participation.
* Active anterior segment ocular disease or using any ocular medication for anterior segment disease (e.g. conjunctivitis, dry-eye disease).
* Current or past condition that might have caused corneal distortion or anterior surface topography abnormalities (e.g. keratoconus, map-dot fingerprint or any other corneal dystrophies, corneal disease or trauma resulting in scarring, pterygium, pellucid marginal degeneration)
* Previous refractive corneal surgery (e.g., laser-assisted in situ keratomileusis (LASIK), photorefractive keratectomy (PRK), corneal transplant, Descemet's Stripping Endothelial Keratoplasty (DSEK) etc.).
* Considered by the Investigator to not be a suitable candidate for participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2018-08-27 (Actual); Study Completion 2018-10-12 (Actual)

PRIMARY OUTCOMES:
Comparison of Through-Focus High Contrast logMAR Visual Acuity for the Test Bifocal Contact Lens Versus that of the Control Bifocal Contact Lens, the Control Single Vision Contact Lens 1, and the Control Single Vision Contact Lens 2 | starting from visit 2 (after enrollment) and finishing with visit 3, the exit visit (up to 60 days after visit 2)
  Visual acuity is measured under high contrast conditions (85% contrast relative to the chart background) at object testing distances of 5.3m, 2m, 1m, 67cm, 50cm and 40cm ("through-focus"), recorded in units of logMAR.

SECONDARY OUTCOMES:
Comparison of Through-Focus Low Contrast logMAR Visual Acuity for the Test Bifocal Contact Lens Versus that of the Control Bifocal Contact Lens, the Control Single Vision Contact Lens 1, and the Control Single Vision Contact Lens 2 | starting from visit 2 (after enrollment) and finishing with visit 3, the exit visit (up to 60 days after visit 2)
  Visual acuity is measured under low contrast conditions (10% contrast relative to the chart background) at object testing distances of 5.3m, 2m, 1m, 67cm, 50cm and 40cm ("through-focus"), recorded in units of logMAR.
Comparison of Visual Quality for the Test Bifocal Contact Lens Versus that of the Control Bifocal Contact Lens, the Control Single Vision Contact Lens 1, and the Control Single Vision Contact Lens 2 | starting from visit 2 (after enrollment) and finishing with visit 3, the exit visit (up to 60 days after visit 2)
  Visual quality is a subjective rating that a participant chooses using an analog rating chart ranging from 0 to 100. Participants are asked to look at the letters that they can read, not the ones that they can't, and rate how sharp those letters are, with 0 denoting "unacceptable" and 100 denoting "excellent." They are asked to reduce their score if any halos, glare, or double vision are present.
Comparison of Fitting Performance for the Test Bifocal Contact Lens Versus that of the Control Bifocal Contact Lens, the Control Single Vision Contact Lens 1, and the Control Single Vision Contact Lens 2 | starting from visit 2 (after enrollment) and finishing with visit 3, the exit visit (up to 60 days after visit 2)
  Fitting performance is measured by visual observation of the contact lens on a participant's eye using a slit lamp biomicroscope and ocular measurement reticle. The position of the lens edge relative to the corneal boundaries both immediately before and immediately after a blink is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Lagana, OD, Principal Investigator
Locations (1):
- Clerio Vision Research Clinic, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ding L, Blackwell R, Kunzler JF, Knox WH. Large refractive index change in silicone-based and non-silicone-based hydrogel polymers induced by femtosecond laser micro-machining. Opt Express. 2006 Nov 27;14(24):11901-9. doi: 10.1364/oe.14.011901. PMID 19529613
- [Background] Ding L, Knox WH, Buhren J, Nagy LJ, Huxlin KR. Intratissue refractive index shaping (IRIS) of the cornea and lens using a low-pulse-energy femtosecond laser oscillator. Invest Ophthalmol Vis Sci. 2008 Dec;49(12):5332-9. doi: 10.1167/iovs.08-1921. Epub 2008 Jul 18. PMID 18641284
- [Background] Xu L, Knox WH, DeMagistris M, Wang N, Huxlin KR. Noninvasive intratissue refractive index shaping (IRIS) of the cornea with blue femtosecond laser light. Invest Ophthalmol Vis Sci. 2011 Oct 17;52(11):8148-55. doi: 10.1167/iovs.11-7323. PMID 21931133
- [Background] Savage DE, Brooks DR, DeMagistris M, Xu L, MacRae S, Ellis JD, Knox WH, Huxlin KR. First demonstration of ocular refractive change using blue-IRIS in live cats. Invest Ophthalmol Vis Sci. 2014 Jul 1;55(7):4603-12. doi: 10.1167/iovs.14-14373. PMID 24985471
- [Background] Wozniak KT, Elkins N, Brooks DR, Savage DE, MacRae S, Ellis JD, Knox WH, Huxlin KR. Contrasting cellular damage after Blue-IRIS and Femto-LASIK in cat cornea. Exp Eye Res. 2017 Dec;165:20-28. doi: 10.1016/j.exer.2017.08.018. Epub 2017 Aug 31. PMID 28866013